CLINICAL TRIAL: NCT01387035
Title: Early Diagnosis of Pulmonary Hypertension in Patients With Inflammatory Rheumatic Connective Tissue Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig, Heidelberg University
Other Study IDs: S-360/2009
Record Dates: First submitted 2011-06-29; First posted 2011-07-04 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Connective Tissue Disease; Pulmonary Hypertension
MeSH Terms: conditions — Connective Tissue Diseases; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purposes of this study are (I), to evaluate various screening methods for their ability to predict and to confirm Pulmonary Hypertension (PH) in scleroderma patients, and (II) to evaluate the incidence of PH (i.e. the number of new cases per year) in scleroderma patients.

ELIGIBILITY:
Inclusion Criteria:

* consent form
* men and women> 18 years
* fulfill the current definition of a collagen vascular disease according to the actual guidelines of the American College of Rheumatology (ACR)

Exclusion Criteria:

* all contraindications for exercise testing
* significant restriction of the left ventricle, unstable coronary artery disease and myocardial infarction in the last 6 months
* patients with other lung diseases (as the pulmonary infestations as part of systemic disease) or related musculoskeletal disorders influencing baseline exercise capacity
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included are all patients who fulfill the current definition of a collagen vascular disease according to the actual guidelines of the American College of Rheumatology (ACR) and who are 18 years or older.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of various screening methods for their ability to predict and to confirm PH in scleroderma patients | 3 years
  Correlate Spiroergometric, lung functional Magnetic Resonance Imaging (MRI) and echocardiographic parameters with invasive hemodynamic findings collected by right heart catheterization: which other non-invasive parameters can be found to detect pulmonary hypertension? Can pulmonary hypertension be detected at rest in the echocardiography? In which patients can only stress-Doppler echocardiography confirm manifest or latent pulmonary hypertension? Is stress-Doppler echocardiography a suitable for early detection of pulmonary hypertension in patients with collagen vascular disease?

SECONDARY OUTCOMES:
Subdivision of patients with connective tissue disease in different degrees of severity | 3 years
  Can spiroergometric findings help to subdivide patients with connective tissue diseases into groups according to degrees of severity, and differ the patients based on spiroergometric findings? To what extent is this distinction comparable with the classifications for the "functional classes" (application for PH according to the New York Heart Association (NYHA) classification)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nagel, MD, Study Director — Center for pulmonary hypertension, Thoraxclinic Heidelberg; Ekkehard Grünig, Professor, Study Director — Center for pulmonary hypertension, Thoraxclinic Heidelberg
Locations (1):
- Center for pulmonary Hypertension, Thoraxclinic Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Nagel C, Marra AM, Benjamin N, Blank N, Cittadini A, Coghlan G, Distler O, Denton CP, Egenlauf B, Fiehn C, Fischer C, Harutyunova S, Hoeper MM, Lorenz HM, Xanthouli P, Bossone E, Grunig E. Reduced Right Ventricular Output Reserve in Patients With Systemic Sclerosis and Mildly Elevated Pulmonary Artery Pressure. Arthritis Rheumatol. 2019 May;71(5):805-816. doi: 10.1002/art.40814. Epub 2019 Apr 10. PMID 30615302
- [Derived] Nagel C, Henn P, Ehlken N, D'Andrea A, Blank N, Bossone E, Bottger A, Fiehn C, Fischer C, Lorenz HM, Stockl F, Grunig E, Egenlauf B. Stress Doppler echocardiography for early detection of systemic sclerosis-associated pulmonary arterial hypertension. Arthritis Res Ther. 2015 Jun 19;17(1):165. doi: 10.1186/s13075-015-0673-7. PMID 26084934